CLINICAL TRIAL: NCT04086043
Title: MultI-eLectrode EndovaScular denervaTiOn in patieNts With Type 2 Diabetes mEllitus (MILESTONE) Study
Brief Title: The MILESTONE Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDNT2DM-2019
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular Denervation (Experimental)
  Interventions: Device: Endovascular Denervation

INTERVENTIONS:
Device: Endovascular Denervation — multi-electrode catheter-based endovascular denervation

SUMMARY:
Sympathetic overactivity induces insulin resistance and type 2 diabetes mellitus (T2DM), so it is assumed that denervation might reduce sympathetic overactivity and improve glucose metabolism and insulin sensitivity. The purpose of this study is to evaluate the effects of multi-electrode catheter-based endovascular denervation on glucose metabolism and insulin sensitivity in patients with T2DM.

DETAILED DESCRIPTION:
Sympathetic overactivity induces insulin resistance and type 2 diabetes mellitus (T2DM), so it is assumed that denervation might improve glucose metabolism and insulin sensitivity. Some clinical studies have shown that glucose metabolism is improved in patients with resistant hypertension both 1 and 3 months after denervation, and fasting glucose, insulin and C-peptide decreased significantly as did insulin resistance assessed by HOMA-IR. But in some clinical studies, denervation did not lead to a significant improvement of insulin sensitivity ≤12 months after treatment, and no effect in systemic sympathetic activity was observed after denervation. Therefore, the efficacy of denervation on glucose metabolism is still in controversy. The investigators wish to investigate the effect of multi-electrode catheter-based endovascular denervation on glucose metabolism and insulin sensitivity in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years and ≤ 70 years old
* Able and willing to provide informed consent
* Patients with established type II diabetes mellitus (HbA1C>7.5%, diet or oral hypoglycaemic agents)
* Clinical stable as demonstrated by no change in background anti-diabetic medication in the last 30 days.
* Anticipated that patients are able to maintain a stable dose of medication for the duration of the study

Exclusion Criteria:

* Arterial anatomy ineligible for endovascular denervation
* History of prior renal artery intervention including balloon angioplasty, stenting or previous renal denervation
* Type 1 diabetes mellitus
* Pregnant, nursing or planning to be pregnant
* Orthostatic hypotension
* eGFR <30 ml/min (MDRD formula)
* Patients that have allergy to contrast agent
* Myocardial infarction, unstable angina pectoris, coronary bypass or percutaneous angioplasty within 3 months before inclusion
* Cerebrovascular accidents and alimentary tract hemorrhage within 3 months before inclusion
* Any medical condition which, in the investigators opinion, may adversely affect the participants safety in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-10 (Estimated); Primary Completion 2022-09-09 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Oral Glucose Tolerance Test from baseline to 6 months | 6 months
  To investigate the influence of endovascular denervation on Oral Glucose Tolerance Test (OGTT).
Changes in glycosylated hemoglobin from baseline to 6 months | 6 months
  To investigate the influence of endovascular denervation on glycosylated hemoglobin (HbA1c).

SECONDARY OUTCOMES:
Changes in Oral Glucose Tolerance Test up to 2 years | 3, 12 and 24 months
  To investigate the influence of endovascular denervation on Oral Glucose Tolerance Test (OGTT).
Changes in glycosylated hemoglobin up to 2 years | 3, 12 and 24 months
  To investigate the influence of endovascular denervation on glycosylated hemoglobin (HbA1c).
Changes in insulin up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of endovascular denervation on insulin.
Changes in catecholamine up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of endovascular denervation on catecholamine.
Changes in glucagon up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of endovascular denervation on glucagon.
Changes in blood pressure up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of endovascular denervation on blood pressure.
Changes in creatinine up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of endovascular denervation on creatinine.
Changes in blood urea nitrogen (BUN) up to 2 years | 3, 6, 12 and 24 months
  To investigate the influence of endovascular denervation on BUN.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No